CLINICAL TRIAL: NCT04027647
Title: A Single-arm, Open-label, Phase 2 Study of Dacomitinib With or Without Dose Titration for the First-line Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer in Subjects With an Epidermal Growth Factor Receptor (EGFR) Activation Mutation
Brief Title: Phase 2 Study of Dacomitinib in NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATORG-003
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: NSCLC Stage IIIB; NSCLC Stage IIIC; NSCLC Stage IV; Recurrent NSCLC; EGFR Positive Non-Small Cell Lung Cancer
Keywords: Stage III NSCLC; Stage IV NSCLC; Vizimpro; EGFR TKI; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Daily administration of oral Dacomitinib
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — 30mg of oral dacomitinib is administered daily for one cycle. After one cycle, a toxicity assessment will be conducted. Subjects will then continue dacomitinib at either 30mg or 45mg.
  Other Names: Vizimpro

SUMMARY:
This is a multi-national, multi-centre, single-arm, open-label, Phase 2 clinical study of the efficacy and safety of first-line treatment with dacomitinib, with or without dose titration, in subjects with newly diagnosed stage IIIB/IIIC/IV or recurrent EGFR-mutation-positive non-small cell lung cancer (NSCLC).

National Cancer Centre Singapore is the lead sponsor acting in a coordinating capacity and the rest of the participating sites are sponsors of their own individual sites.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a voluntarily given, personally signed and dated, written informed consent document;
* Male or female adult as defined by local regulation;
* The presence of an EGFR activating mutation (exon 19 deletion or the L858R mutation in exon 21) in tumor specimen determined by the local laboratory;
* Evidence of newly diagnosed stage IIIB/IIIC/IV (based on Union for International Cancer Control (UICC) staging system version 8) or recurrent (minimum of 12 months disease free interval between completion of systemic therapy and recurrence of NSCLC required) NSCLC of adenocarcinoma histo- and/or cytopathology or its pathologically accepted variants using tumor specimen (assessed according to accepted standards by a local laboratory). For this purpose the World Health Organization/International Association of Study of Lung Cancer Histologic Classification of Lung Cancer Criteria will be used and the diagnosis of NSCLC NOS (not otherwise specified), squamous or mixed adeno-squamous lung carcinomas will not be allowed;
* Have an ECOG PS of 0 or 1;
* No prior treatment with systemic therapy for locally advanced or metastatic NSCLC. Completed neoadjuvant/adjuvant chemotherapy/immunotherapy and/or combined modality chemotherapy/radiation therapy permitted only in cases in which there is a minimum of 12 months disease free interval between completion of systemic therapy and recurrence of NSCLC. Prior treatment with a EGFR-TKI or other TKIs is not allowed;
* Radiologically measurable disease by RECIST v1.1 criteria:

  1. At least one target lesion that has not previously been radiated, and is measurable according to RECIST v1.1;
  2. Acceptable radiologic procedures for disease assessment include contrast enhanced conventional or spiral computed tomography (CT), or contrast enhanced magnetic resonance imaging (MRI); Non-contrast CT scan is acceptable only for subjects who are both allergic to intravenous contrast and unable to cooperate with MRI, or MRI is not available. The following are not allowed as sole documentation of target lesions: CT component of positron emission tomography (PET)/CT, ultrasound alone, nuclear scans (including bone or PET scans), chest X-ray or bone radiographs, and tumor markers;
* Adequate organ function, including:

  1. Estimated creatinine clearance ≥30 mL/min (as determined by Cockcroft-Gault formula or the study site's standard formula);
  2. Absolute neutrophil count (ANC) ≥1500 cells/mm3;
  3. Platelets ≥100,000 cells/mm3;
  4. Hemoglobin ≥10.0 g/dL;
  5. Bilirubin ≤1.5 x ULN;
  6. AST (also known as SGOT) and ALT (also known as SGPT) ≤2.5 x ULN (≤5.0 x ULN if hepatic metastases).
* Female subjects must be postmenopausal (defined as 12 months of amenorrhea following last menses), or they or their partners must be surgically sterile, or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the investigator using following criteria:

  a. Acceptable contraception for women include implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), sexual abstinence, or a partner who has been surgically sterile (e.g. by vasectomy) for at least 6 months. Acceptable contraception for a male includes surgical sterility (e.g. by vasectomy) for at least 6 months, sexual abstinence, or condoms plus spermicide.
* All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to starting study treatment;
* Male subjects or their female partners must be surgically sterile or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter. The definition of effective contraception will be based on the judgment of the investigator. Or female partners must be postmenopausal (defined as 12 months of amenorrhea following last menses);
* Willing and able to comply with study scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any evidence of mixed histo- and/or cytology that includes elements of small cell or carcinoid lung cancer. Variations of adenocarcinoma are allowed, however no squamous element can be present;
* An EGFR exon 20 T790M or exon 20 insertion mutation;
* Symptomatic brain or leptomeningeal metastases, who are neurologically unstable or require increasing doses of steroids and/or anti-seizure medications to manage CNS symptoms within two weeks prior to starting dacomitinib;
* Any previous anti-cancer systemic treatment of locally advanced, or metastatic NSCLC including but not limited to chemotherapy, targeted therapies, small molecules, EGFR-TKIs and other TKIs, monoclonal antibodies, anti-cancer vaccines, immunotherapy, radiotherapy (other than palliative radiotherapy to lesions that will not be followed for tumor assessment on this study, i.e., non-target lesions). Completed neoadjuvant/adjuvant chemotherapy/immunotherapy and/or combined modality chemotherapy/ radiation therapy permitted only in cases in which there is a minimum of 12 months disease free interval between completion of systemic therapy and recurrence of NSCLC. Prior treatment with a EGFR-TKI or other TKIs is not allowed;
* Any surgery (not including minor procedures such as lymph node biopsy), palliative radiotherapy or pleurodesis within 2 weeks of baseline assessments;
* Any clinically significant gastrointestinal abnormalities that may impair intake, transit or absorption of the study drug, such as the inability to take oral medication;
* Current enrollment in another therapeutic clinical study;
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this study; or known drug abuse/alcohol abuse;
* History of, or currently suspected, diffuse non-infectious pneumonitis or interstitial lung disease including:

  1. Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease;
  2. Pre-existing idiopathic pulmonary fibrosis evidenced by CT scan at baseline;
  3. Insufficient lung function as determined by either clinical examination or an arterial oxygen tension of <70 Torr.
* Any history of rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
* Clinically important abnormalities in cardiac rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, second degree heart block, third degree heart block) OR:

  1. Diagnosed or suspected congenital long QT syndrome;
  2. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
  3. Prolonged QTc interval on ECG; QTc must be less than CTCAE v5.0 Grade 2 (≤480 msec) using Fridericia's or Bazett's correction formula with a manual reading by the investigator if required. The ECG may be repeated for evaluation of eligibility after management of correctable causes for observed QTc prolongation;
  4. Any history of second or third degree heart block;
  5. Heart rate <45 beats per minute on ECG in the presence of clinical symptoms (e.g., hypotension, evidence of hypoperfusion);
* Severely impaired (defined as Child-Pugh Class C) hepatic dysfunction;
* Prior malignancy: Subjects will not be eligible if they have history of, or evidence of active disease of another concurrent malignancy within the previous five years. Exception would be effectively treated past history of non-melanoma skin cancer or in-situ cervical cancer with no evidence of active disease;
* Other severe acute or chronic medical condition that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study;
* Use of CYP2D6 substrates where minimal increases in concentration of the CYP2D6 substrate may lead to serious or life-threatening toxicities, including but not limited to procainamide, pimozide, and thioridazine from screening to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment to the date of disease progression or death due to any cause at 12 months
  Percentage of subjects with PFS at 12 months

SECONDARY OUTCOMES:
Overall Survival | From the start of treatment to the date of death for any cause, up to 3 years
Objective Response Rate | From the start of treatment until disease progression, up to 3 years
  Proportion of subjects with a best overall response of either complete response (CR) or partial response (PR)
Time to Treatment Failure | From the start of treatment to the last dose of treatment, up to 3 years
Intracranial Objective Response Rate | From the start of treatment until disease progression, up to 3 years
  Proportion of subjects with a best overall response of either CR or PR of intracranial disease
Intracranial Progression-Free Survival | From the start of treatment to the date of intracranial progression or death due to any cause, up to 3 years
Number of incidences of adverse events | From start of treatment to 28 days after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tan, BSc, MBBS, PhD, Principal Investigator — National Cancer Centre Singapore (Lead Sponsor)
Locations (9):
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Malaysia (3):
  - Sarawak General Hospital, Kuching, Sarawak
  - University Malaya Medical Centre, Kuala Lumpur
  - Beacon Hospital, Petaling Jaya
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (2):
  - Dong-A University Hospital, Busan
  - Seoul National University Hospital, Seoul
- Thailand (2):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok